CLINICAL TRIAL: NCT07116954
Title: Root Resorption and Alveolar Bone Changes in the Maxillary Canine Retraction Using Ni Ti Closed-coil Springs Versus Elastomeric Chains (A Split -Mouth Cone Beam CT Study)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Hassan Mahdy, Principal Investigator (Postgraduate Researcher in Orthodontics), Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Ethical committee
Record Dates: First submitted 2025-07-15; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Orthodontic Patients Indicated for Upper First Premolar Extraction; Orthodontic Patients Indicated for Maxillary Canine Retraction
Keywords: Niti coil springs; Canine Retraction; Elastomeric Chains; Root resorption; CBCT
MeSH Terms: conditions — Root Resorption

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1: Elastomeric chains will be used on the right side, and NiTi closed-coil springs will be use (Experimental)
  Interventions: Procedure: Twenty-Two adult Patients who indicated for bilateral maxillary first premolar extraction will be randomly assigned into two equal group.; Procedure: Canin retraction with NiTi Closed-Coil Springs and elastomeric chains
- Group2: NiTi closed-coil springs will be used on the right side, Elastomeric chains will be used on (Experimental)
  Interventions: Procedure: Canin retraction with NiTi Closed-Coil Springs and elastomeric chains

INTERVENTIONS:
Procedure: Twenty-Two adult Patients who indicated for bilateral maxillary first premolar extraction will be randomly assigned into two equal group. — Group1: Elastomeric chains will be used on the right side, and NiTi closed-coil springs will be used on the left side. Group2: NiTi closed-coil springs will be used on the right side, Elastomeric chains will be used on the left side.
  Arms: Group1: Elastomeric chains will be used on the right side, and NiTi closed-coil springs will be use
Procedure: Canin retraction with NiTi Closed-Coil Springs and elastomeric chains — Comparison between canine retraction using NiTi closed-coil springs versus elastomeric chains

SUMMARY:
This study will be carried out to asses root resorption and alveolar bone changes in the maxillary canine retraction using NiTi closed-coil springs versus elastomeric chains with cone beam CT

ELIGIBILITY:
* Inclusion Criteria:

  * Patients aged 16 years or older
  * Patients indicated for fixed orthodontic appliances
  * Patients indicated for bilateral extraction of maxillary first premolars
  * Patients who have not undergone any previous orthodontic treatment
* Exclusion Criteria:

  * Patients with a history of craniofacial trauma, anomalies, or congenital defects
  * Patients currently taking anticoagulant drugs affecting bone metabolism
  * Patients with a history of trauma or pathology involving the maxillary canines
  * Patients with periodontally compromised teeth

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change in Apical Root Length After Canine Retraction | Baseline (prior to canine retraction) and 6 months after retraction
  Measurement of apical root length (in millimeters) using CBCT images at T1 and T2 to assess root resorption on both retraction methods.
Change in Alveolar Bone Thickness After Canine Retraction | Baseline (prior to canine retraction) and 6 months after retraction
  Quantitative measurement of alveolar bone thickness (in millimeters) using CBCT images taken at baseline (T1) and post-treatment (T2) in both NiTi closed-coil spring and elastomeric chain sides.

SECONDARY OUTCOMES:
Change in Probing Depth | Baseline and 6 months post-treatment
  Measurement of probing depth (in millimeters) on both sides at baseline and 6 months
Change in Plaque Index | Baseline and 6 months post-treatment
  Scoring of plaque accumulation using the Silness-Löe Plaque Index (score range: 0 to 3; higher score = worse outcome)
Change in Bleeding Index | Baseline and 6 months post-treatment
  Evaluation using the Gingival Bleeding Index (score range: 0 to 3; higher score = worse outcome)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD), including CBCT-based measurements of alveolar bone height and root resorption, will be shared. Data will be available beginning 6 months after study completion via a secure external repository (link will be provided in the References section). Access will be granted to researchers upon request and subject to approval.
Supporting Information: Study Protocol, SAP, CSR